CLINICAL TRIAL: NCT03219112
Title: Training Balance Control Using Virtual Reality Games in Children With Cerebral Palsy and Typically Developing Children
Brief Title: Training Balance Control in Children With Cerebral Palsy Using Virtual Reality Games
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B670201525057; 2015/0666 (Other: Commission medical ethics University Hospital Ghent)
Record Dates: First submitted 2017-02-17; First posted 2017-07-17 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Cerebral Palsy, Spastic
Keywords: balance; rehabilitation; exergaming; virtual reality
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 15 cp children + 10 typically developing children (anticipated) Will have 8 weeks VR training Will have 1 VR training session
  Interventions: Other: Balance rehabilitation using X-box One & Kinect
- Control (No Intervention): 15 cp children (anticipated) Will not have 8 weeks of VR training Will not have 1 VR training session

INTERVENTIONS:
Other: Balance rehabilitation using X-box One & Kinect — the virtual reality games (Kinect sports rivals) can be controlled with movements of the body that are registered through the kinect camera.
  Arms: Intervention

SUMMARY:
In this study the clinical relevance of the use of commercially available virtual reality games in the rehabilitation of balance will be assessed in children with cerebral palsy. It will be investigated how different commercially available platforms (i.e. Xbox One + Kinect and Nintendo Wii + balance board) will affect the compensations of children with cerebral palsy to preserve their balance. The effect of 1 training session will be assessed as well as the effect of a long-term training of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. children diagnosed with cerebral palsy (spastic type)
2. age: 8-11 years and 11 months
3. bilateral CP (diplegia) & unilateral CP (hemiplegia)
4. GMFCS level 1 & 2
5. able to independently stand still for 2 minutes
6. sufficient cooperation to participate in the measurements and training

Exclusion Criteria:

1. No informed consent
2. surgery of the lower limbs that affects mobility
3. Botulinum-toxin A treatment within 6 months prior to inclusion in the study
4. vestibular deficits, benign vertigo, ADHD or instable epilepsia

For typically developing children:

Inclusion criteria;

1. age: 8-11 years and 11 months
2. no history of neurologic, musculoskeletal or other impairments that could affect mobility

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-08-25; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Pediatric Balance Scale compared to baseline | measured at baseline, after 40 minutes (of training), and after 8 weeks of training
  Clinical balance scale with 14 items such as standing unsupported for 30 sec.

SECONDARY OUTCOMES:
Change in Bruininks-Oseretsky test for motor proficiency - subscale 'balance' and 'speed & agility' compared to baseline | measured at baseline, after 40 minutes (of training), and after 8 weeks of training
  Subscales of a clinical balance scale
Change in Upper body kinematics compared to baseline | measured at baseline, after 40 minutes (of training), and after 8 weeks of training
  Trunk and arm movements measured using 3d movement registration
Change in Posturography compared to baseline | measured at baseline, after 40 minutes (of training), and after 8 weeks of training
  Measurements on a moveable force-platform including the limits of stability during standing

CONTACTS AND LOCATIONS:
Locations (1):
- Vakgroep REVAKI (Ghent University - Ghent University hospital), Ghent, Belgium

REFERENCES:
- [Derived] Meyns P, Blanckaert I, Bras C, Jacobs N, Harlaar J, van de Pol L, Plasschaert F, Van Waelvelde H, Buizer AI. Exergaming improves balance in children with spastic cerebral palsy with low balance performance: results from a multicenter controlled trial. Disabil Rehabil. 2022 Oct;44(20):5990-5999. doi: 10.1080/09638288.2021.1954704. Epub 2021 Aug 9. PMID 34365883